CLINICAL TRIAL: NCT03247309
Title: Phase 1 Study Evaluating Genetically Modified Autologous T Cells Expressing a T-cell Receptor Recognizing a Cancer/Germline Antigen in Patients With Recurrent and/or Refractory Solid Tumors (ACTengine® IMA201-101)
Brief Title: TCR-engineered T Cells in Solid Tumors (ACTengine IMA201-101)
Acronym: ACTengine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immatics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMA201-101
Record Dates: First submitted 2017-08-01; First posted 2017-08-11 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor; Cancer; Recurrent Solid Tumors; Refractory Solid Tumors
Keywords: T-cell therapy; immunotherapy; adoptive cellular therapy; T-Cell Receptor; IMA201; Cytotherapy; Cell Therapy; Gene Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- IMA201 Product (Experimental): * Pre-conditioning by non-myeloablative chemotherapy with Fludarabine and Cyclophosphamide
  * One dose of IMA201 product will be infused intravenously. Up to four dose levels will be evaluated. At least two patients per cohort will be treated.
  * Post-infusion of IMA201 product, administration of low-dose recombinant human interleukin-2
  Interventions: Biological: IMA201 Product; Diagnostic Test: IMADetect®

INTERVENTIONS:
Biological: IMA201 Product — The cell dose will be based on viable CD3+CD8+ HLA-Dextramer+ cells per body surface area (BSA) as defined by the Mosteller formula.
Diagnostic Test: IMADetect® — IMADetect® is developed as a companion diagnostic to aid in selecting patients with relapsed and/or refractory solid cancers who might be eligible for enrollment in clinical trials with investigational IMA201 therapy. IMADetect® is intended for investigational use only.

SUMMARY:
The study purpose is to establish the safety and tolerability of IMA201 in patients with solid tumors that express melanoma-associated antigen 4 and/or 8 (MAGEA4/8).

DETAILED DESCRIPTION:
SCREENING: Patient eligibility will be determined by HLA (human leukocyte antigen) screening and the biomarkers screening. If the patient is eligible, white blood cells will be taken during leukapheresis for the manufacture of the IMA201 product.

MANUFACTURING: IMA201 product will be made from the patient's white blood cells.

TREATMENT: Lymphodepletion with cyclophosphamide and fludarabine will occur in the days before the IMA201 infusion to improve the duration of time that IMA201 stays in the body.

After IMA201 infusion, a low dose of IL-2 will be given twice daily for a period of time.

Patients will be closely monitored for safety and for a total of 3 years post IMA201 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Pathologically confirmed advanced and/or metastatic solid tumor
* Patients may enter screening procedure before, during, or after the last available indicated standard of care treatment. There is no limitation for prior anti cancer treatments.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* HLA phenotype positive for the study
* Patients must have measurable disease according to RECIST 1.1
* Disease accessible to biopsy
* Adequate pulmonary function per protocol
* Adequate organ and bone marrow function per protocol
* Acceptable coagulation status per protocol
* Adequate hepatic function per protocol
* Adequate renal function per protocol
* Patient's tumor must express tumor antigen by qPCR using a fresh tumor biopsy specimen
* Life expectancy more than 3 months
* Confirmed availability of production capacities for IMA201 product
* Patients must have recurrent/progressing and/or refractory solid tumors and must have received or not be eligible for all available indicated standard of care treatment.
* For hepatocellular carcinoma (HCC) patients only, Child-Pugh score of ≤ 6
* IMA201 product must have passed all of the release tests
* Female patient of childbearing potential must use adequate contraception prior to study entry until 12 months after the infusion of IMA201
* Male patient must agree to use effective contraception or be abstinent while on study and for 6 months after the infusion of IMA201
* The patient must have recovered from any side effects of prior therapy to Grade 1 or lower (except for non-clinically significant toxicities; e.g., alopecia, vitiligo) prior to lymphodepletion. As determined by the investigator, the patient may still be eligible if the patient has not fully recovered from Grade ≥ 2 toxicities if these toxicities are not anticipated to further improve (e.g., chronic neuropathy) and such toxicities are not anticipated to worsen with the lymphodepletion therapy

Exclusion Criteria:

* History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years
* Solid tumors with low likelihood of tumor biomarker expression per protocol
* Pregnant or breastfeeding
* Serious autoimmune disease Note: At the discretion of the investigator, these patients may be included if their disease is well controlled without the use of immunosuppressive agents.
* History of cardiac conditions as per protocol
* Prior stem cell transplantation or solid organ transplantation
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study
* History of hypersensitivity to cyclophosphamide (CY), fludarabine (FLU), or IL-2, or to any of the rescue medications
* History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician
* HIV infection, active hepatitis B virus (HBV), active hepatitis C virus (HCV) infection, ongoing active anti-HCV treatment or detectable HBV or HCV viral load at the most recent laboratory report. Patients with both HBV and HCV infections will be excluded from screening

  1. Patients with a history of HCV infection and with an undetectable viral load per the most recent laboratory report and/or completed anti-HCV treatment but are HCV antibody positive are permitted.
  2. History of treated HBV infection is permitted if the viral load is undetectable per the most recent laboratory report. Note: HCC patients with controlled HBV infection, as defined by resolved (anti-hepatitis B surface antigen [HBs-Ag] antibody (Ab) negative, anti-core antigen [HBc Ag] Ab positive) or chronic stable (anti HBs-Ag Ab positive) HBV infection will be eligible for screening. Patients with active HBV infection who are not on anti-HBV treatment will be excluded.
* Any condition contraindicating leukapheresis, lymphodepletion, low-dose IL-2, and/or IMA201 treatment
* Patients with any active viral infection
* Patients with active brain metastases

NOTE: Patients with a history of brain metastases may be eligible, if an imaging scan with contrast enhancement not older than 4 weeks is able to exclude the existence of currently active brain metastasis, and steroid therapy has been discontinued for ≥2 weeks.

* Treatment with protocol-defined excluded treatments, medical devices, and/or procedures per protocol
* Concurrent participation in an interventional part of another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | up to 3 years post-treatment
Determination of the maximum tolerated dose (MTD) | until 21 days post treatment

SECONDARY OUTCOMES:
Duration of infused T cells over time (Persistence of T cells) | up to 3 years post-treatment
Tumor response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 and immune-related RECIST (irRECIST) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cedrik Britten, MD, PhD, Study Director — Immatics US, Inc.
Locations (5):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (3):
  - Universitätsklinikum Bonn, Venusberg-Campus 1, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Fetscherstr. 74, Dresden, Saxony
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fritsche J, Rakitsch B, Hoffgaard F, Romer M, Schuster H, Kowalewski DJ, Priemer M, Stos-Zweifel V, Horzer H, Satelli A, Sonntag A, Goldfinger V, Song C, Mahr A, Ott M, Schoor O, Weinschenk T. Translating Immunopeptidomics to Immunotherapy-Decision-Making for Patient and Personalized Target Selection. Proteomics. 2018 Jun;18(12):e1700284. doi: 10.1002/pmic.201700284. Epub 2018 Apr 10. PMID 29505699